CLINICAL TRIAL: NCT04191291
Title: Time for Lunch: The Impact of Lunch Time Constraints on Child Eating Behaviors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 19412
Record Dates: First submitted 2019-06-13; First posted 2019-12-09 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Time Constraints During School Meals

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shortened lunch period (Experimental): The amount of seated lunch time will be 10 minutes.
  Interventions: Behavioral: Lunch period length
- Longer lunch period (Experimental): The amount of seated lunch time will be 20 minutes.
  Interventions: Behavioral: Lunch period length

INTERVENTIONS:
Behavioral: Lunch period length — We are randomly allocating a 10 minute or 20 period of seated lunch time.

SUMMARY:
Recent peer-reviewed observational evidence suggests that school children receive anywhere from 10-33 minutes of seated lunch time and that students with less time to eat discard higher amounts of milk, entrée (i.e. protein items), grains, and vegetables. This waste is a missed nutritional and food security opportunity and also negatively impacts the environment. The purpose of this study is to estimate the impact that lunch time constraints have on child food selection, consumption and waste behaviors using a crossover trial design, where the duration of seated lunch times are randomly allocated to be either 10 minutes or 20 minutes each day.

ELIGIBILITY:
Inclusion Criteria:

* Must be enrolled in local summer camp

Exclusion Criteria:

* None

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
Food item selection | Ranges from 5 days to 20 days, depending upon how long each participant elects to enroll in the summer camp
  The type and number of school meal components selected by students to eat for lunch.
Food item consumption | Ranges from 5 days to 20 days, depending upon how long each participant elects to enroll in the summer camp
  The weight of each school meal component that was consumed by each child during lunch. Each measured in grams.
Food item waste | Ranges from 5 days to 20 days, depending upon how long each participant elects to enroll in the summer camp
  The weight of each school meal component that was discarded by each child during lunch. Each measured in grams.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Burg X, Metcalfe JJ, Ellison B, Prescott MP. Effects of Longer Seated Lunch Time on Food Consumption and Waste in Elementary and Middle School-age Children: A Randomized Clinical Trial. JAMA Netw Open. 2021 Jun 1;4(6):e2114148. doi: 10.1001/jamanetworkopen.2021.14148. PMID 34156451